CLINICAL TRIAL: NCT04555902
Title: Evaluation of Postcard Mailers Enhanced With Behavioral Nudges to Promote Mammogram Screening
Brief Title: Evaluation of Mailers Promoting Mammogram Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Screening
Other Study IDs: 2020-0761
Record Dates: First submitted 2020-09-04; First posted 2020-09-21 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Mass Screening; Communication; Mammography; Risk Reduction Behavior; Economics, Behavioral; Psychology; Loss Frame; Fear Appeals; Reciprocity
MeSH Terms: conditions — Breast Neoplasms; Communication; Risk Reduction Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: 1 x 3 design
Who Masked: Participant, Care Provider
Masking Description: Participants and providers are not aware of the different mailer versions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Mailer and Small Gift (Active Comparator): A postcard encourages mammograms and includes a small gift.
  Interventions: Behavioral: Postcard; Behavioral: Small Gift
- Mailer with Loss Frame, Risks, and Small Gift (Experimental): The postcard is enhanced with language that further emphasizes the risks but also clearly describes how early detection with a test can reduce those risks; a small gift is included.
  Interventions: Behavioral: Postcard; Behavioral: Small Gift; Behavioral: Loss Frame and Fear Appeals
- Mailer with Loss Frame, Risks, and No Gift (Experimental): The postcard is enhanced with language that further emphasizes the risks but also clearly describes how early detection with a test can reduce those risks; the small gift is not included.
  Interventions: Behavioral: Postcard; Behavioral: Loss Frame and Fear Appeals

INTERVENTIONS:
Behavioral: Postcard — The postcard includes appeals to get annual mammograms and provides information for ordering a mammogram.
Behavioral: Small Gift — Pink socks are included in the mailer. The gift increases salience of the mailer and it potentially promotes reciprocation from the recipient in the form of ordering a mammogram.
  Arms: Mailer with Loss Frame, Risks, and Small Gift; Standard Mailer and Small Gift
Behavioral: Loss Frame and Fear Appeals — The postcard is enhanced with language that frames the situation in terms of losses. It also uses fear appeals by stating the risks of breast cancer, while also stating that a mammogram screening is an accessible way to address those risks.
  Arms: Mailer with Loss Frame, Risks, and No Gift; Mailer with Loss Frame, Risks, and Small Gift

SUMMARY:
In this evaluation, 3 different versions of mailers promoting annual mammograms are being sent to women on the month of their 50th and 64th birthdays. The researchers hypothesize that the use of behavioral nudges in the mailers should lead to increased uptake in mammogram screening.

DETAILED DESCRIPTION:
Mammogram screening for women, starting at age 50, can significantly reduce the risk of complications due to breast cancer. As part of an existing outreach campaign, the health system mails a postcard and small gift (pink socks) to women on the month of their 50th and 64th birthdays to promote annual mammogram screening.

The researchers are evaluating two new versions of the mailers against a standard mailer to see which version leads to greater uptake in mammograms. The new mailers have content that applies behavioral nudge theory - specifically, loss frames and fear appeals - to encourage taking action. One of the two new versions does not include the small gift, to test whether its inclusion or exclusion has any effect on mammogram screening.

ELIGIBILITY:
Inclusion Criteria:

* Female Geisinger Health Plan members turning 50 and 64 in that month
* For the 2020 campaign, birthdays from June 2020 (as opposed to August 2020) will be included due to a temporary suspension of the outreach program due to the COVID-19 pandemic since June
* For the pre-post examination of the 2019 campaign, all months in that year will be included

Exclusion Criteria:

- Members who are on the do not contact list at Geisinger Health Plan

Ages: 50 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1342 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Mammogram Completion at 6 months (2020) | 6 months from intervention start date
  Binary variable indicating whether a mammogram was completed

SECONDARY OUTCOMES:
Mammogram Completion at 12 months (2020) | 12 months from intervention start date
  Binary variable indicating whether a mammogram was completed (a longer time frame allows for late responses)
Primary Care Provider Visits at 6 months (2020) | 6 months from intervention start date
  Number of visits (proxy for increased preventative health care)
Primary Care Provider Visits at 12 months (2020) | 12 months from intervention start date
  Number of visits (proxy for increased preventative health care)
Obstetrician-Gynecologist Visits at 6 months (2020) | 6 months from intervention start date
  Number of visits (proxy for increased preventative health care)
Obstetrician-Gynecologist Visits at 12 months (2020) | 12 months from intervention start date
  Number of visits (proxy for increased preventative health care)
Breast Cancer Diagnosis at 6 months (2020) | 6 months from intervention start date
  Binary variable indicating whether the recipient was diagnosed with breast cancer
Breast Cancer Diagnosis at 12 months (2020) | 12 months from intervention start date
  Binary variable indicating whether the recipient was diagnosed with breast cancer
Emergency Department Visits at 6 months (2020) | 6 months from intervention start date
  Number of Emergency Department Visits (proxy for increased costly utilization of health system resources)
Emergency Department Visits at 12 months (2020) | 12 months from intervention start date
  Number of Emergency Department Visits (proxy for increased costly utilization of health system resources)

OTHER OUTCOMES:
Mammogram Completion at 12 months (2019) | 12 months from 2019 intervention start date
  Binary variable indicating whether a mammogram was completed to be used for exploratory pre-post comparisons
Primary Care Provider Visits at 12 months (2019) | 12 months from 2019 intervention start date
  Number of visits to be used for exploratory pre-post comparisons (proxy for increased preventative health care)
Breast Cancer Diagnosis at 12 months (2019) | 12 months from 2019 intervention start date
  Binary variable indicating whether the woman was diagnosed with breast cancer
Emergency Department Visits at 12 months (2019) | 12 months from 2019 intervention start date
  Number of Emergency Department Visits (proxy for increased costly utilization of health system resources)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings. The PI did not examine or analyze any data from this study prior to this registration.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT04555902/Prot_SAP_000.pdf